CLINICAL TRIAL: NCT03538652
Title: Just-In-Time Adaptive Interventions for Addictive Behaviors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to the 2020 pandemic
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 999918095; 18-DA-N095
Record Dates: First submitted 2018-05-25; First posted 2018-05-29 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Addiction
Keywords: cognitive-behavioral therapy (CBT); Mindfulness; Opiates; Ecological Monetary Assessment (EMA); Microrandomized Trial
MeSH Terms: conditions — Behavior, Addictive | interventions — Cognitive Behavioral Therapy; Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1, Arm 1: Formative Interviews (Placebo Comparator): Outpatient adults who are in treatment for opioid use disorder (OUD) participate in a formative-interview phase (one hour) to drive intervention formation for the trial participants groups.
  Interventions: Other: Formative Interviews (not an intervention)
- Phase 2, Arm 1: Just-in-time adaptive intervention (JITAI) group (Experimental): Outpatient adults who are in treatment for opioid use disorder (OUD) will receive electronic messages on their smartphone via an app and education on some basic principles of CBT and ACT. Participants will designate four one-hour time bands within their typical waking hours, covering morning through late evening. During each of those time bands, the app will push a pair of assessments, given 20 minutes apart.
  Interventions: Behavioral: Cognitive-behavioral therapy (CBT); Behavioral: Acceptance and commitment therapy (ACT)
- Phase 2, Arm 2: Ecological momentary assessment (EMA) group (control group) (Active Comparator): Outpatient adults who are in treatment for opioid use disorder (OUD) will receive electronic messages on their smartphone via an app. Participants will designate four one-hour time bands within their typical waking hours, covering morning through late evening. During each of those time bands, the app will push a pair of assessments, given 20 minutes apart.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Formative Interviews (not an intervention) — One hour formative-interview session
  Arms: Phase 1, Arm 1: Formative Interviews
Behavioral: Cognitive-behavioral therapy (CBT) — In CBT, negative emotional states are viewed as problems to be solved, and the client learns skills to solve them.
  Arms: Phase 2, Arm 1: Just-in-time adaptive intervention (JITAI) group
Behavioral: Acceptance and commitment therapy (ACT) — In ACT, negative emotional states are viewed as a necessary and potentially valuable component of a full life. When they occur, the goal is not to solve them, but to experience them in an observant, curious, nonjudgmental way-a practice referred to as mindfulness.
  Arms: Phase 2, Arm 1: Just-in-time adaptive intervention (JITAI) group
Other: No intervention — Control group with no intervention administered
  Arms: Phase 2, Arm 2: Ecological momentary assessment (EMA) group (control group)

SUMMARY:
Background:

Many smartphone apps intend to help people with addictions. But not enough is known about how they should work. Researchers want to study an app that gives people the advice they need, just when they need it. This is a Just-In-Time Adaptive Intervention (JITAI). To create a good JITAI, researchers need to know what approaches work best at different moments.

Objective:

To develop ways to treat addiction with a smartphone app.

Eligibility:

Adults ages 18-75 who use heroin or other opioids

Design:

Participants will be screened in another protocol.

Participants will visit a Baltimore clinic 3 days a week to give urine and breath samples.

Some participants will get their treatment at this clinic.

Participants will answer questions about their personality and stress.

Participants will randomly be assigned to the JITAI group or a comparison group.

Participants will have a training session on using the smartphone app. JITAI participants will also watch a video about the written messages they will see in the app.

Weeks 3-10: Participants will carry a smartphone. Four times a day, it will beep and ask questions. These will be about the participants' activities and mood. The JITAI group will see a short message after. The message is meant to be helpful.

For the first 16 evenings, JITAI participants will get more information on the phone.

Answers to the app's questions will be transferred automatically from the smartphone to secure computers at the NIH.

During the last week, participants can choose the kind of messages they see.

Week 11: participants will return the smartphone and answer questions.

Weeks 12-16, participants who are getting their medicine from the research clinic will be encouraged to transfer to other clinics. Otherwise, they will have their dose slowly reduced to zero.

DETAILED DESCRIPTION:
BACKGROUND: Our research group has made extensive use of ecological momentary assessment (EMA) to understand people's daily experiences with opioid craving, use, and lapse. We have also administered clinic-based psychotherapies such as cognitive-behavioral therapy (CBT), in which clients learn to avoid, escape, resolve, or reframe problems (such as stress) that can trigger lapses to drug use. CBT contrasts with ACT (Acceptance and Commitment Therapy), a mindfulness-based approach in which difficult thoughts and feelings are viewed as necessary and potentially valuable components of a full life, to be experienced observantly rather than resolved or reframed. CBT and ACT can and do coexist in a single treatment plan, but we know of no systematic attempt to reconcile their differences. We have also not tried to administer either of them on a mobile device.

OBJECTIVE: To test a just-in-time adaptive intervention (JITAI)-a treatment given when and where it is needed. Our JITAI will be delivered via smartphone app and will combine elements of two widely used treatments for addiction: CBT and ACT. Our goal is not to bring another branded app onto the market, but rather to clarify when and for whom the generic components of such apps are effective or not. This will include determining when CBT is more helpful than ACT and vice versa.

PARTICIPANT POPULATION: Outpatient adults who are physically dependent on opioids - up to 185 enrolled (35 for a formative-interview phase, 150 for a trial) for a target of 115 evaluable (30 interviewees, 85 trial participants). Target enrollment will include 40% women and 60% minorities (mostly African-American). In the trial, some participants will receive buprenorphine in our clinic, and others will be receiving buprenorphine or methadone elsewhere; this is a procedural matter, not a component of the experimental design.

EXPERIMENTAL DESIGN: After a formative-interview phase, the study will be run as a microrandomized trial that will also include a conventionally randomized between-groups clinical-trial component. In microrandomization, interventions are randomized at the momentary level within person; the effect is measured proximally (e.g., 20 minutes later). This is a powerful way to assess the effects of different interventions administered in the field and to examine strategy-situation fit, i.e., whether interventions are differentially effective under specific momentary circumstances. We are powering our study mostly to detect

* (1) any effect of CBT or ACT versus control moments with no intervention given, and
* (2) preferential advantages of CBT over ACT, and vice versa, as a function of the participant's ability to control (change, escape) a given situation.

The between-groups aspect of the design (JITAI group versus EMA-only control group) is needed to demonstrate an effect of our JITAI on traditional, distal measures of outcome, such as reductions in opioid use.

METHODS: In the formative-interview phase, we will conduct interviews with people in treatment for OUD who express interest in using a mobile treatment app. We will ask them about day-to-day challenges they currently face in maintaining progress toward their treatment goals, and ask them what might be helpful. Then we will show them item lists, onscreen mockups, and/or functional demos, and we will ask interviewees to comment on the app's likely usefulness, its likely pitfalls, and how we could improve it.

In the clinical trial, participants will be randomized to one of two groups (JITAI vs. EMA-only control).

* During weeks 1-2, all participants will have baseline assessments of coping styles and personality, and all JITAI participants will be shown a video introducing basic concepts of CBT and ACT.
* For weeks 3-10 (8 weeks), participants will carry smartphones for EMA with or without JITAI.
* During week 11, participants will be readministered some of the assessments from baseline.

Participants receiving buprenorphine from us will then be offered a dose taper or encouraged to transfer to continued treatment elsewhere. All participants will come to our clinic thrice weekly for urine testing throughout participation.

PRIMARY OUTCOME MEASURES:

1. Proximal effects of CBT and ACT messages in the JITAI group: decreases over 20-minute intervals in craving and negative mood, with increases in self-efficacy
2. strategy-situation fit in the JITAI group
3. group differences in distal effects of treatment (week 11 versus week 2) in terms of self-efficacy and coping flexibility

SECONDARY OUTCOME MEASURES:

1. Trait predictors of differential responses to CBT and ACT, in the JITAI group
2. group differences in frequency of opioid-positive urine over time
3. time courses of responsiveness to ACT vs. CBT, in the JITAI group
4. whether the intervention types that benefit participants most when pushed by the app are the same ones participants choose when subsequently given the opportunity to pull interventions.

ELIGIBILITY:
* INCLUSION CRITERIA:

Phase 1: Formative interviews.

The enrollment ceiling is 35 outpatients (to collect evaluable data from 30) who meet these criteria: (1) Age 18-75; (2) physical dependence on opioids (by self-report); (3) interest in receiving the types of treatment about which we will be conducting interviews.

Phase 2: Clinical trial with microrandomization.

The enrollment ceiling is 150 outpatients (to collect evaluable data from 85, of whom 50 will be randomized to JITAI, and 35 to EMA control). Treatment may be provided by us in the form of office-based buprenorphine treatment (OBOT) or may be provided elsewhere (Treatment Elsewhere, TE).

Participants must meet these criteria:

OBOT participants: (1) Age 18-75; (2) physical dependence on opioids (by positive urine and/or frank opioid withdrawal); (3) interest in receiving the types of treatment we are testing.

Treatment Elsewhere (TE) participants: (1) Age 18-75; (2) receiving methadone or buprenorphine treatment for opioid dependence from a qualified provider in the community; (3) interest in receiving the types of treatment we are testing.

EXCLUSION CRITERIA:

Phase 1: Formative interviews. (1) cognitive impairment severe enough to preclude informed consent or valid interview responses.

Phase 2: Clinical trial with microrandomization.

OBOT participants:

* (1) History of any DSM-V psychotic disorder; history of bipolar disorder; current Major Depressive Disorder;
* (2) unresolved symptoms of PTSD that, in the investigators view, would make it risky for the participant to undertake mindfulness exercises (e.g., observing all one's current negative thoughts and emotions) in an unsupervised setting;
* (3) current dependence on alcohol or sedative-hypnotic, e.g. benzodiazepine (by DSM-V criteria);
* (4) cognitive impairment severe enough to preclude informed consent or valid self-report;
* (5) Any condition that interferes with urine collection;
* (6) medical illness (e.g., cirrhosis, nephritic syndrome, thyroid disease, ischemic heart disease, epilepsy, adrenal insufficiency, etc.) or medications that, in the view of the investigators, would compromise participation in research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Epstein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Some health information collected may be placed into one or more scientific databases after it has been stripped of identifiers such as name, address or account number, so that it may be used for future research on any topic and shared broadly for research purposes. A researcher who wants to study the information must apply to the database and be approved.
Access Criteria: We will share some protocol data with our scientific research partners inside or outside the NIH. Research partners outside the NIH sign an agreement with the NIH to share data. This agreement indicates the type of data that can be shared and what can be done with those data.

RESULTS

PARTICIPANT FLOW:
Period: Phase 1
Arm/Group | Phase 1, Arm 1: Formative Interviews | Phase 2, Arm 1: Just-in-time Adaptive Intervention (JITAI) Group | Phase 2, Arm 2: Ecological Momentary Assessment (EMA) Group (Control Group)
Started | 9 | 0 | 0
Completed | 9 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1, Arm 1: Formative Interviews | Phase 2, Arm 1: Just-in-time Adaptive Intervention (JITAI) Group | Phase 2, Arm 2: Ecological Momentary Assessment (EMA) Group (Control Group)
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phase 1, Arm 1: Formative Interviews
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Opioid Craving Rating
Description: Change in opioid craving within 20 minutes from receiving app messages. Participants designates four one-hour time bands within their typical waking hours, covering morning through late evening. During each of those time bands, the app will push a pair of assessments, given 20 minutes apart. Pre and post assessment ratings will be done using rating scale on the app from 0 to 100 ("0 = not at all" to "100- as much as possible"). Higher number indicates more opioid craving. Participants will complete ratings four times daily for 11 weeks. Analysis will be done in multilevel models.
Time Frame: Within 20 minutes from receiving app message
Population: Per protocol document, outcome analysis applies only to the Just-in-time adaptive intervention (JITAI) group. Study was closed before any data were collected for the primary outcomes.
Arm/Group | Phase 2, Arm 1: Just-in-time Adaptive Intervention (JITAI) Group
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Mood Rating
Description: Change in mood within 20 minutes from receiving app message. Rating will be done using rating scale on the app from 0 to 100 ("0 = not at all" to "100 = as much as possible"). Higher number indicates more negative mood. Participants will complete ratings four times daily for 11 weeks. Analysis will be done in multilevel models.
Time Frame: Within 20 minutes from receiving app message
Population: as for outcome 1
Arm/Group | Phase 2, Arm 1: Just-in-time Adaptive Intervention (JITAI) Group
Number analyzed (Participants) | 0

3. Primary Outcome: Change in Self-efficacy
Description: Change in self-efficacy within 20 minutes from receiving app message. Rating will be done using rating scale on the app from 0 to 100 ("0 = not at all" to "100 = as much as possible"). Higher number indicates more positive self-efficacy. Participants will complete ratings four times daily for 11 weeks. Analysis will be done in multilevel models.
Time Frame: Within 20 minutes from receiving app message
Population: as for outcome 1
Arm/Group | Phase 2, Arm 1: Just-in-time Adaptive Intervention (JITAI) Group
Number analyzed (Participants) | 0

4. Primary Outcome: Strategy-situation Fit of Cognitive-behavioral Therapy (CBT)
Description: The analysis will be a test of whether cognitive-behavioral therapy (CBT) messages are most effective in controllable situations and Acceptance and Commitment Therapy (ACT) messages are most effective in noncontrollable situations. A situation will be categorized as noncontrollable when a participant gives a response of less than 50/100 on either of these two "pre" items: (1) "I could easily be somewhere else right now if I wanted," (2) "I could easily get out of what I'm doing right now." Otherwise, will categorize the situation as controllable. Analysis will be done in multilevel models.
Time Frame: Within 20 minutes from receiving app message
Population: as for outcome 1
Arm/Group | Phase 2, Arm 1: Just-in-time Adaptive Intervention (JITAI) Group
Number analyzed (Participants) | 0

5. Primary Outcome: Strategy-situation Fit of Acceptance and Commitment Therapy (ACT)
Description: as for outcome 4
Time Frame: Within 20 minutes from receiving app message
Population: as for outcome 1
Arm/Group | Phase 2, Arm 1: Just-in-time Adaptive Intervention (JITAI) Group
Number analyzed (Participants) | 0

6. Primary Outcome: Change in Coping Self-efficacy
Description: Participants coping self-efficacy will be assessed using the Drug-Taking Confidence Questionnaire (DTCQ-8), an 8-item measure of coping self-efficacy in the context of resisting lapses to drug misuse and administered by clinician. Each item is scored from 0 to 100. Higher score indicates more confidence. Assessment will be administered at weeks 2 and 11. Data will be analyzed via analysis of covariance (ANCOVA), with score from week 2 as the covariate to assess change (change = week 11 minus week 2).
Time Frame: week 2 versus week 11
Population: Study was closed before any data were collected for the primary outcomes.
Arm/Group | Phase 2, Arm 1: Just-in-time Adaptive Intervention (JITAI) Group | Phase 2, Arm 2: Ecological Momentary Assessment (EMA) Group (Control Group)
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Change in Coping-style Flexibility
Description: Coping-style flexibility was assessed using the Coping Orientation to Problems Experienced (COPE) questionnaire, a 60-item self-report scale assessing both general coping styles and coping behaviors in specific situations. Each item is rated 1 = I usually don't do this at all, to 4 = I usually do this a lot, with total score of 60 to 240. Higher score indicates improved coping. Assessment will be administered at weeks 2 and 11. Data will be analyzed via analysis of covariance (ANCOVA), with score from week 2 as the covariate to assess change (change = week 11 minus week 2).
Time Frame: week 2 versus week 11
Population: Study was closed before any data were collected for the primary outcomes.
Arm/Group | Phase 2, Arm 1: Just-in-time Adaptive Intervention (JITAI) Group | Phase 2, Arm 2: Ecological Momentary Assessment (EMA) Group (Control Group)
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Change in Flexibility Index Test (FIT)
Description: The Flexibility Index Test (FIT-60), a standard measure of traits associated with mindfulness, such as "I observe my feelings without losing myself in them" and "It is OK if I remember something unpleasant," and (reverse scored) "I believe that some of my thoughts are abnormal or bad and that I shouldn't think like that." Each item is rated 0 (completely disagree) to 6 (completely agree) for total score of 0 to 360. Higher score indicates better psychological flexibility. Assessment will be administered at weeks 2 and 11. Data will be analyzed via analysis of covariance (ANCOVA), with score from week 2 as the covariate to assess change (change = week 11 minus week 2).
Time Frame: week 2 versus week 11
Population: Study was closed before any data were collected for the primary outcomes.
Arm/Group | Phase 2, Arm 1: Just-in-time Adaptive Intervention (JITAI) Group | Phase 2, Arm 2: Ecological Momentary Assessment (EMA) Group (Control Group)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: One day for participants in the formative interview (phase 1)
Arm/Group | Phase 1, Arm 1: Formative Interviews
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
Study was closed before any data were collected for the primary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT03538652/Prot_SAP_000.pdf